CLINICAL TRIAL: NCT06282172
Title: Effect of Treatment With BTL-785F Device on Submental Subcutaneous Adipose Tissue - Histological Evaluation
Brief Title: Histological Evaluation of BTL-785F Device's Effect on Submental Subcutaneous Adipose Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTL-785_CTUS1600
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2024-02

CONDITIONS: Fat Burn
Keywords: submentum; fat reduction; adipocyte; apoptosis; double chin
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment with BTL-785-7 (Experimental): Active treatment with BTL-785-7
  Interventions: Device: Treatment with BTL-785-7
- Control (No Intervention): No active treatment

INTERVENTIONS:
Device: Treatment with BTL-785-7 — Treatment with BTL-785-7 delivering simultaneously radiofrequency (RF) and HIFES energy on the submental area
  Arms: Treatment with BTL-785-7

SUMMARY:
This study aims to evaluate the safety and effectiveness of the BTL-785F system equipped with the BTL-785-7 applicator for non-invasive reduction of subcutaneous submental fat.

DETAILED DESCRIPTION:
This study aims to evaluate the safety and effectiveness of the BTL-785F system equipped with the BTL-785-7 applicator for non-invasive reduction of subcutaneous submental fat. The changes in the fat tissue related to the morphology (shape, size and count) will be assessed histologically. The presence of biochemical apoptotic indicators will be analysed in the adipocytes.

The study is a prospective single-center open-label two-arm study. The subjects will be enrolled and assigned into two study groups; Group A which will receive active treatment (5 subjects) and Group B (2 subjects), will serve as the control, and will not receive any treatment to verify the treatment outcomes.

Subjects will be required to complete one (1) treatment visit and three (3) follow-up visits (at 24 hours, 7 days and 14 days post treatment). The third follow-up visit is for safety evaluation.

At baseline inclusion and exclusion criteria will be verified upon obtaining informed consent from the patient.

Punch biopsies (3mm diameter) will be obtained from the treatment area for histologic analysis. In the control group, biopsy will be obtained from the location corresponding to the treatment area in the active group.

Safety measures will include documentation of adverse events (AE) during and after the treatment procedures and at the follow up visits and if needed medical assistance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects over 21 years of age seeking treatment for reduction of submental fat
* Subjects should be able understand the investigative nature of the treatment, the possible benefits and side effects, and must sign the Informed Consent Form
* Presence of clearly visible excess fat in submentum as deemed appropriate by the Investigator
* Subjects willing and able to abstain from partaking in any facial treatments other than the study procedure during study participation
* Willingness to comply with study instructions, to return to the clinic for the required visits, and to undergo punch biopsy of the submental area

Exclusion Criteria:

* Local bacterial or viral infection in the area to be treated
* Local acute inflammation in the area to be treated
* Impaired immune system caused by any immunosuppressive illness, disease or medication
* Isotretinoin and tretinoin-containing medication use in the past 12 months
* Skin related autoimmune diseases
* Radiation therapy and/or chemotherapy
* Poor healing and unhealed wounds in the treatment area
* Metal implants
* Permanent implant in the treated area
* Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body
* Facial dermabrasion, facial resurfacing, or deep chemical peeling in the treatment area within 3 months prior to the treatment
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
* History of skin disorders, keloids, abnormal wound healing and dry or fragile skin
* History of any type of cancer
* Active collagen diseases
* Cardiovascular diseases (such as vascular diseases, peripheral arterial disease, thrombophlebitis, hypersensitive carotid sinus and thrombosis)
* Pregnancy/nursing or IVF procedure
* History of bleeding coagulopathies, use of anticoagulants
* Any active condition in the treatment area, such as sores, psoriasis, eczema, rash and rosacea
* Any surgical procedure in the treatment area within the last three months or before complete healing
* Poorly controlled endocrine disorders, such as diabetes
* Acute neuralgia and neuropathy
* Kidney or liver failure
* Nerve insensitivity (sensitivity disorders) to heat in the treatment area
* Varicose veins, pronounced edemas
* Prior use of dermal fillers, botulinum toxin, lasers, etc. therapies in the treated area that can influence the study results at the investigator discretion
* Unwillingness/inability to not change their usual cosmetics and especially not to use fat reduction, anti-aging or anti-wrinkles products in the treated area during the duration of the study including the follow-up period
* Electroanalgesia without exact diagnosis of pain etiology
* Neurological disorders (such as multiple cerebrospinal sclerosis, epilepsy)
* Blood vessels and lymphatic vessels inflammation
* Any other disease or condition at the investigator discretion that may pose risk to the patient or compromise the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Investigation of the effects of the BTL-785F device (with BTL-785-7 applicator) on the morphology of submental adipose cells. | 6 months
  Histological evaluation of changes in the shape and size of submental adipose cells, based on biopsies obtained from both the treatment and control groups.

SECONDARY OUTCOMES:
Investigation of post-treatment adipocyte apoptosis | 6 months
  Histologically analyze the adipocyte tissue for the change in apoptosis markers (caspase-3/7 and Bcl-2) levels.
Incidence of Treatment-related Adverse Events | 6 months
  Evaluation of the safety of the BTL-785F device with BTL-785-7 applicator for non-invasive treatment of the submental area throught monitoring of adverse events
Comfort Evaluation Assessed by Therapy Comfort Questionnaire | 6 months
  Evaluation of therapy comfort using the 5-point Likert scale Therapy Comfort Questionnaire given to subjects after the treatment, where the best possible answer would be "strongly agree" and the worst "strongly disagree". The questionnaire includes pain sensation rating on the scale from 0 (no pain) to 10 (worst possible pain), where 0 (no pain) represents the best possible outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Schweiger Dermatology PC, Research Division, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldberg DJ. Adipocyte Apoptosis Following a Novel Method for Double Chin Reduction: A Pilot Human Histology Study. J Cosmet Dermatol. 2025 Jan;24(1):e16643. doi: 10.1111/jocd.16643. Epub 2024 Nov 13. PMID 39536780